CLINICAL TRIAL: NCT01492491
Title: Collaborative Study on Outcome of Antioxidant Vitamines, Microinflammation Parameters and Middle-high Toxins in ESRD Patients Treated With Online HDF, HFR and SUPRA-HFR
Brief Title: Collaborative Research on HFR High Flux
Acronym: SALATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Sanitaria Locale di Cagliari (Other)
Collaborators: Bellco s.r.l. (Unknown); Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Piergiorgio Bolasco, Head Physician, Azienda Sanitaria Locale di Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRC-01; ASLCagliariPBolascosolismo52 (Registry Identifier: 231152PBolasco)
Record Dates: First submitted 2011-12-10; First posted 2011-12-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Inflammation
Keywords: SUPRA-HFR; adsorpition; vitamins; large toxins
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard HFR therapy (No Intervention): standard HFR hemodiafiltration therapy
- SUPRA-HFR therapy (Active Comparator): SUPRA-HFR hemodiafiltration therapy
  Interventions: Device: SUPRA-HFR

INTERVENTIONS:
Device: SUPRA-HFR — usual dialytic prescription for duration, frequency, acid buffer and anticoagulation regimen.
  Arms: SUPRA-HFR therapy

SUMMARY:
The purpose of this study is to evaluate the serum concentrations of antoxidant vitamines A, C, E, inflammatory cytokines and middle-large toxins in patients treated with online hemodiafiltration, standard HFR and SUPRA-HFR.

DETAILED DESCRIPTION:
Today, as the research work of EUTOX group highlights, large cytokines and protein-bound solutes are gaining a relevant attention because of their emerging role as mortality predictors.

Online hemodiafiltration (online HDF) has demonstrated to offer a significant depuration for small and middle toxins, but removal of protein-bound solutes is scarce. Synthetic high-flux membranes do not allow infact significant removal of molecules heavier than 15-20 KDa. Super-flux membranes may enhance online HDF convective transport but it would surely expose the patient to unacceptable losses of albumin, vitamines and aminoacids because of the non selectivity of the convective transport.

HFR is a renal replacement therapy that utilizes convection, diffusion and adsorption. It uses a double-stage filter that consists of a high-flux polyethersulfone hemofilter in the first convective stage and a low-flux polyethersulfone filter in the second diffusive stage. The stages of the filter allow complete separation of convection from diffusion. The convective part of the first stage allows pure ultrafiltrate (UF) to pass through a sorbent resin cartridge. The first convective/adsorption stage has no net fluid removal. The blood and reinfused clean UF then undergo traditional dialysis. The second stage works by classicaHD and in this final stage the weight loss occurs. HFR has demonstrated in various clinical trials to reduce the microinflammatory state with no albumin loss and minimal aminoacids losses, thanks to the high selectivity of the resin sorbent.

SUPRA-HFR is a newly developed HDF therapy based on the HFR concept scheme, which includes a super-flux membrane in the first section, coupled with an empowered resin sorbent. This should significantly enhance large solutes depuration, overcoming online HDF flaws.

Therefore we proposed a prospective, multicenter, randomized study comparing online HDF, standard HFR and SUPRA-HFR. After a wash-out stabilization period of 4 months in post-dilution online HDF, an expected number of 50 patients will be randomized either in standard HFR (25) or in SUPRA-HFR (25) and followed for 6 months. Primary end points focus on the the removal of protein-bound solutes, inflammation and nutritional state. In addition, ESAs doses and hemoglobin levels will be assessed and compared between treatment groups.

This study will provide strong evidence on the safe and clinically effective use of super-flux membranes, introduced with SUPRA-HFR therapy. It is highly likely that the outcomes of this study will affect the daily clinical practice of Italian and European dialysis centers because of the potential innovation brought to the market.

The following hypotheses will be tested:

* SUPRA-HFR selectivity will reduce consistently the albumin, aminoacids and vitamines A, C, E losses compared to online HDF.
* SUPRA-HFR better preservation of the nutritional parameters, coupled with the possibility to remove protein-bound toxins and cytokines should lead to a higher reduction of the microinflammatory status, compared to online HDF and to standard HFR.
* SUPRA-HFR impact on inflammation status should ameliorate the anemia management by reducing the administered ESAs doses.

ELIGIBILITY:
Inclusion Criteria:

* dialysis vintage > 6 months
* well functioning vascular access (QB > 300 mL/min)
* informed consent given

Exclusion Criteria:

* polycystic kidney disease (PKD)
* significant acute or chronic inflammatory comorbidities
* non-renal related anemia
* blood transfusions in the last 2 months before enrollment
* alcohol or drugs abuse
* malignant neoplasm
* hemoglobinopathy or myelopathy
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
selective depuration of large uraemic toxins and reduction of nutrient losses | 1 year
  evaluation of the serum level of albumin, antioxidant vitamins and cytokines (IL6, IL1-beta)

SECONDARY OUTCOMES:
amelioration of the anemia management | 1 year
  evaluation of ESAs dose, Hb level

CONTACTS AND LOCATIONS:
Overall Officials: Piergiorgio Bolasco, MD, Principal Investigator — Azienda Sanitaria Locale di Cagliari
Locations (11):
- Italy (11):
  - Territorial dialysis service, Regional Health system nephrology and dialysis department, Cagliari
  - Nephrology and dialysis, SS. Trinità Hospital, Cagliari
  - Nephrology and dialysis, Civil Hospital, La Maddalena
  - Nephrology and dialysis, Civil Hospital, Lanusei
  - Nephrology and dialysis department, Versilia Hospital, Lido di Camaiore
  - Nephrology and dialysis department, Civil Hospital, Macomer
  - Nephrology and dialysis, San Francesco Hospital, Nuoro
  - Nephrology and dialysis, San Martino Hospital, Oristano
  - Nephrology and dialysis department, Bonaria Hospital, San Gavino Monreale
  - Nephrology and dialysis, San Camillo Hospital, Sorgono
  - Nephrology and dialysis, Dettori Hospital, Tempio

REFERENCES:
- [Background] Wratten ML, Ghezzi PM. Hemodiafiltration with endogenous reinfusion. Contrib Nephrol. 2007;158:94-102. doi: 10.1159/000107239. PMID 17684347
- [Background] Bolasco PG, Ghezzi PM, Serra A, Corazza L, Murtas S, Mascia M, Cossu M, Ferrara R, Cogoni G, Cadinu F, Casu D, Contu B, Passaghe M, Ghisu T, Ganadu M, Logias F. Hemodiafiltration with endogenous reinfusion with and without acetate-free dialysis solutions: effect on ESA requirement. Blood Purif. 2011;31(4):235-42. doi: 10.1159/000322400. Epub 2011 Jan 14. PMID 21242676
- [Background] Panichi V, Manca-Rizza G, Paoletti S, Taccola D, Consani C, Filippi C, Mantuano E, Sidoti A, Grazi G, Antonelli A, Angelini D, Petrone I, Mura C, Tolaini P, Saloi F, Ghezzi PM, Barsotti G, Palla R. Effects on inflammatory and nutritional markers of haemodiafiltration with online regeneration of ultrafiltrate (HFR) vs online haemodiafiltration: a cross-over randomized multicentre trial. Nephrol Dial Transplant. 2006 Mar;21(3):756-62. doi: 10.1093/ndt/gfi189. Epub 2005 Nov 22. PMID 16303780
- [Derived] Palleschi S, Ghezzi PM, Palladino G, Rossi B, Ganadu M, Casu D, Cossu M, Mattana G, Pinna AM, Contu B, Ghisu T, Monni A, Gazzanelli L, Mereu MC, Logias F, Passaghe M, Amore A, Bolasco P; Sardinian Study Group. Vitamins (A, C and E) and oxidative status of hemodialysis patients treated with HFR and HFR-Supra. BMC Nephrol. 2016 Aug 26;17(1):120. doi: 10.1186/s12882-016-0315-6. PMID 27566671